CLINICAL TRIAL: NCT04682288
Title: An Interventional, Open Label, Non-randomized, Phase Ia Safety and Tolerability Study of Levofloxacin Ocular Implant in Subjects Undergoing Routine Cataract Surgery.
Brief Title: Levofloxacin Ocular Implant for Ocular Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PolyActiva Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEVO-CS101
Record Dates: First submitted 2020-11-08; First posted 2020-12-23 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levofloxacin Ocular Implant (Experimental): Biphasic levofloxacin antibiotic implant
  Interventions: Drug: Levofloxacin Ocular Implant

INTERVENTIONS:
Drug: Levofloxacin Ocular Implant — Levofloxacin Ocular Implant an implant that delivers a bolus dose of levofloxacin and a constant daily dose for a further 5-7 days.

SUMMARY:
This is a multi center, open label, interventional study in one eye of 5 subjects scheduled for uncomplicated cataract surgery with administration of a single Levofloxacin Ocular Implant in the posterior sulcus of the surgical eye at the end of cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cataract in the intent to treat eye
* Endothelial cell density in the study eye of at least 2000 cells per mm2

Exclusion Criteria:

* history of ocular inflammation including, macular degeneration, uveitis, macular edema or corneal edema
* recent surgery in the study eye
* subjects receiving a glaucoma device in conjunction with cataract surgery
* subjects with a compromised posterior capsule during surgery
* corneal disease that prevents effective imaging of endothelium including Fuch's Dystrophy.
* sensitivity to fluoroquinolones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Ocular Inflammation | 90 days
  Change assessed according to Standardization of Uveitis Nomenclature (SUN) Grading Scale
Endothelial Cell Density | 90 days
  Change in number of central corneal endothelial cells per mm2
Intraocular Pressure (IOP) | 90 days
  Change in IOP measured by Goldmann applenation tonometry

SECONDARY OUTCOMES:
Administration procedure | 1 week
  Number of actuation's required to expel implant

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gira, MD, Principal Investigator — Opthalmology Consultants Ltd
Locations (3):
- United States (2):
  - Ophthalmology Consultants Ltd, St Louis, Missouri
  - Carolina Cataract and Laser Centre, Ladson, South Carolina
- Melbourne Eye Specialists, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No